CLINICAL TRIAL: NCT05361473
Title: Evaluation of a Mattress With Phase Change Material Can be Helpful to Start Hypothermia During Transport Before Admissions to Neonatal Ward
Brief Title: Evaluation of a PCM Mattress to Treat HIE Infants During Transport
Acronym: PCMhypo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: National Children's Hospital, Vietnam (Other); Calmark Sweden AB (Unknown)
Responsible Party: Principal Investigator, Linus Olson, Project Investigator, Dr., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PCMcooling test study Vietnam
Record Dates: First submitted 2020-09-11; First posted 2022-05-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Newborn Hypoxic-Ischemic Encephalopathy
Keywords: Asfyxia; HIE; Infections; Lactate dehydrogenase
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The NeoHilda Point of care method (Active Comparator): Evaluating baby including lactate dehydregenase Levels measured in umbilical core blood using the fast point of care method called Neo Hilda
  Interventions: Device: The NeoHilda Point of care method
- No Measurement of LDH (Sham Comparator): Evaluating baby without Lactate dehydrogenase result
  Interventions: Procedure: Traditional evaluation

INTERVENTIONS:
Device: The NeoHilda Point of care method — This is a procedure that measures Lactate dehydrogenase in a fast and reliable way from only 10 microliter of blood. Using a small point of care card and a Smartphone for analysis.
  Other Names: Neo Hilda, Calmark Sweden AB
  Arms: The NeoHilda Point of care method
Procedure: Traditional evaluation — Traditional way of evaluation
  Arms: No Measurement of LDH

SUMMARY:
Background the research proposed herein is in line with the Swedish Research Council's current focus on International collaborations and postdoctoral work abroad. In this case the child brain and translational and clinical infant brain research. Neonatal hypoxic ischemic encephalopathy in term infants constitutes a serious health problem, not the least due to its often life-long consequences in the form of cerebral palsy and other forms of brain dysfunction.

An estimated 3-5 of every 1000 live term births are affected, a quarter of which with severe symptoms; 10-30% of the affected children do not survive, 30% suffer life-long disabilities. The incidence may be 10-fold higher in the developing world. In Sweden, an estimated 200 children are born each year with hypoxic ischemic asphyxia or oxygen deprivation during delivery of a severity necessitating treatment, in order to reduce future handicap. Not only the brain, but also other organs, such as the heart, liver or kidney can be damaged by hypoxic ischemia.

In clinical trials, proof has been obtained that cooling can have positive effects counteracting brain injury induced by oxygen deprivation (asphyxia). Recent research suggests that cooling may also have a positive effect in stroke during the pre-treatment/transportation to hospital phase.

PCM. A material with phase change properties (PCM) can be a chemical element, a solution or a substance with high melting energy. It melts/solidifies at a precise temperature and can store considerable amounts of energy (heat) before changing from one phase to another. The study group have used elements or solutions that change between solid and fluid phases within a narrow temperature interval. The most common use of PCM today is for energy storage, accomplished by having the PCM change between solid and fluid phases. Phase changes that include other PCMs, high temperatures and/or gas phases are less useful in medical applications due to the need of either large volumes in a low pressure setting or smaller amounts in a high pressure setting, increasing the risk for mistakes or secondary injury to medical staff or patients. For the clinical purposes of hypothermic treatment described here, the Glauber salt-based PCM in a mattress form developed by the applicant has near ideal properties; it is completely safe, does not cause over-cooling, can be reused many times, eliminates cooling fluctuations, is easy to handle and biodegradable.

DETAILED DESCRIPTION:
Background. The research proposed herein, is in line with the Swedish Research Council's current focus on International collaborations and postdoctoral work abroad. In this case the child brain and translational and clinical infant brain research. Neonatal hypoxic ischemic encephalopathy in term infants constitutes a serious health problem, not the least due to its often life-long consequences in the form of cerebral palsy and other forms of brain dysfunction.

An estimated 3-5 of every 1000 live term births are affected, a quarter of which with severe symptoms; 10-30% of the affected children do not survive, 30% suffer life-long disabilities [1-9]. The incidence may be 10-fold higher in the developing world. In Sweden, an estimated 200 children are born each year with hypoxic ischemic asphyxia or oxygen deprivation during delivery of a severity necessitating treatment, in order to reduce future handicap. Not only the brain, but also other organs, such as the heart, liver or kidney can be damaged by hypoxic ischemia.

In clinical trials, proof has been obtained that cooling can have positive effects counteracting brain injury induced by oxygen deprivation (asphyxia) [1-7, 9]. Recent research suggests that cooling may also have a positive effect in stroke (30000 new cases/year in Sweden) during the pre-treatment/transportation to hospital phase.

PCM. A material with phase change properties (PCM) can be a chemical element, a solution or a substance with high melting energy [10-13]. It melts/solidifies at a precise temperature and can store considerable amounts of energy (heat) before changing from one phase to another. The study project have used elements or solutions that change between solid and fluid phases within a narrow temperature interval. The most common use of PCM today is for energy storage, accomplished by having the PCM change between solid and fluid phases. Phase changes that include other PCMs, high temperatures and/or gas phases are less useful in medical applications due to the need of either large volumes in a low pressure setting or smaller amounts in a high pressure setting, increasing the risk for mistakes or secondary injury to medical staff or patients. For the clinical purposes of hypothermic treatment described here, the Glauber salt-based PCM in a mattress form developed by the applicant has near ideal properties; it is completely safe, does not cause over-cooling, can be reused many times, eliminates cooling fluctuations, is easy to handle and biodegradable. III. Methods Whole body cooling with PCM mattresses is straightforward. Rectal temperature will be monitored in standard ways. Several other vital parameters, such as LDH in blood, and standard procedures will be used to monitor condition of the infants continuously. 15 days after treatment, MRI will be carried out at the National Hospital of Pediatrics in Hanoi. Follow up of the treated and control children will be carried out at 18 months of age and will be the bases of the final evaluation of the clinical trial.

Design. The project is based on the applicant's dual expertise in engineering and medicine. The applicant developed a key technology, cooling using a special PCM composition, recently. The applicant has also participated in multicenter hypothermia studies of newborn infants (including the TOBY trial). As part of the PhD program, the applicant has also participated in animal research using a large newborn anesthetized piglet therapeutic hypothermia model in collaboration with Dr. Nicola Robertson and her team at University College of London. These experiences enable design of the current project.

Assessment is done continuously during the first 60 minutes. If criteria A and B are fulfilled, treatment is started before 6 hours of life. Amplitude-integrated EEG is not mandatory to start hypothermia treatment. V. Significance The significance of the research project would be to demonstrate that a novel PCM-technology based method, previously not clinically tested, and could be developed all the way to clinical implementation. In infants, the method has the specific advantage of being easily applied already during transport to a hospital, which makes it possible to begin cooling of many children within the current 6 hr. age limit. If hypoxic ischemic encephalopathy can be prevent fully or partly by hypothermia with PCM, major life-long health improvements for many children worldwide, would result. PCM-based cooling is safe, simple, reusable, environmentally safe, non-toxic, and independent of clean water and electricity and a method where the risk of temperature undershooting causing additional damage is eliminated.

ELIGIBILITY:
Inclusion Criteria:

All children admitted to the neonatal ward above 32w of age, considered for blood sampling.

Exclusion Criteria:

* parental consent missing
* Gestational age less than 33 weeks postnatal age or above 36 hours after birth

Max Age: 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2013-08; Primary Completion 2024-08-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient classification/ window of oppertunity Hypothermia during transport or start late | At 96 hours after admission to study for each patient, During the data collection time of the study.
  Efficacy of sending patient to right level of care. Is it better to start early during transport by using the PCM mattress or miss the window of opportunity of 6h due to long transportation and/or long decision making. Usage of questionnaire that collect outcome of hypothermia.

OTHER OUTCOMES:
Feasibility and validation of the HildaNeo method, usage. | Each case is evaluated immediately after the intervention/procedure but the results of all combined is evaluated after completion of study to avoid bias.
  Did the HildaNeo and the LDH value ( in 4 segments) help improve care for patients.
  The feasibility of the HildaNeo card is evaluated for each patient by their Responsible doctor after use of card, using a questionnaire checking if the doctor felt better and more sure of how to classify the patient for hypothermia treatment and start cooling or not after have seen the LDH result diveded into 4 segments; No value recorded/low value, normal, high, and extreem high LDH value. The Question are answered Yes or No.
LDH as indicator for HIE | From date of sample taken during the study until end of data collection, max 100 month. Each case is evaluated immediately after the intervention/procedure but the results of all combined is evaluated after completion of study to avoid bias.
  Does the LDH test (Hilda Neo) detect infants at high risk for HIE in the group admitted before 6 hours of age.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Lagercrantz, Professor, Study Director — Karolinska Institutet; Khu TK Dung, Prof, Vdir., Principal Investigator — National Hospital of Pediatrics
Locations (1):
- Neonatal unit, National hospital of Pedriatrics, Hanoi, Dong Da, Vietnam

REFERENCES:
- [Background] Karlsson M, Dung KT, Thi TL, Borgstrom E, Jonstam K, Kasstrom L, Winbladh B. Lactate dehydrogenase as an indicator of severe illness in neonatal intensive care patients: a longitudinal cohort study. Acta Paediatr. 2012 Dec;101(12):1225-31. doi: 10.1111/apa.12014. PMID 22963670
- [Background] Karlsson M, Wiberg-Itzel E, Chakkarapani E, Blennow M, Winbladh B, Thoresen M. Lactate dehydrogenase predicts hypoxic ischaemic encephalopathy in newborn infants: a preliminary study. Acta Paediatr. 2010 Aug;99(8):1139-44. doi: 10.1111/j.1651-2227.2010.01802.x. Epub 2010 Mar 19. PMID 20236255
- [Background] Wiberg-Itzel E, Akerud H, Andolf E, Hellstrom-Westas L, Winbladh B, Wennerholm UB. Association between adverse neonatal outcome and lactate concentration in amniotic fluid. Obstet Gynecol. 2011 Jul;118(1):135-142. doi: 10.1097/AOG.0b013e318220c0d4. PMID 21691171
- [Background] Thoresen M, Liu X, Jary S, Brown E, Sabir H, Stone J, Cowan F, Karlsson M. Lactate dehydrogenase in hypothermia-treated newborn infants with hypoxic-ischaemic encephalopathy. Acta Paediatr. 2012 Oct;101(10):1038-44. doi: 10.1111/j.1651-2227.2012.02778.x. Epub 2012 Jul 27. PMID 22775455
- [Derived] Tran HTT, Tran DM, Le HT, Hellstrom-Westas L, Alfven T, Olson L. Cooling during transportation of newborns with hypoxic ischemic encephalopathy using phase change material mattresses in low-resource settings: a randomized controlled trial in Hanoi, Vietnam. BMC Pediatr. 2024 Aug 8;24(1):509. doi: 10.1186/s12887-024-04987-6. PMID 39118070